CLINICAL TRIAL: NCT00970645
Title: A Prospective Multicenter Study Comparing Endobronchial and Endoscopic Ultrasound-Guided FNA to Mediastinoscopy/Thoracoscopy in the Staging and Early Detection of Metastases in Lung Cancer
Brief Title: Study Comparing EBUS & EUS to Mediastinoscopy in Staging and Detection of Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar study published results
Sponsor: Mayo Clinic (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Eric S. Edell, M.D., Mayo Clinic, Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-002240; DOD protocol A-12345.8
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; mediastinum; endobronchial ultrasound fine needle aspiration; endoscopic ultrasound; mediastinoscopy; surgical or minimally invasive evaluation of mediastinum; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Mediastinoscopy; Thoracoscopy; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- traditional mediastinoscopy/thoracoscopy (Active Comparator): Traditional Mediastinoscopy used to detect or stage lung cancers.
  Interventions: Procedure: Mediastinoscopy/thoracoscopy
- EBUS/EUS (Active Comparator): Minimal invasive technique for staging/detecting lung cancer.
  Interventions: Procedure: EBUS/EUS

INTERVENTIONS:
Procedure: Mediastinoscopy/thoracoscopy — Mediastinoscopy used to detect/stage lung cancer.
  Other Names: Lung biopsy
  Arms: traditional mediastinoscopy/thoracoscopy
Procedure: EBUS/EUS — Minimal invasive technique to stage/detect lung cancer.
  Other Names: Endobronchial Ultrasound; Endoscopic Ultrasound
  Arms: EBUS/EUS

SUMMARY:
This is a prospective randomized clinical trial with the study cohort comprised of all male and female patients over the age of 21 presenting to the study site for evaluation of lung cancer. The study will enroll 300 subjects, with 150 in each arm. Three sites will be in the study, Mayo Rochester, Mayo Jacksonville and Medical University of South Carolina. Mayo Rochester will enroll approximately 125 subjects. This study does not require subjects to undergo any additional procedures than what they would receive per standard medical care. The consenting subjects will receive EUS and /or EBUS- guided FNA or Mediastinoscopy/Thoracoscopy.

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial of males and females age 21 or older being evaluated for lung cancer. The study will enroll approximately 300 subjects (150 in each arm) at 3 participating centers (MUSC, Mayo Clinic Rochester and Jacksonville). This sample size will provide sufficient statistical power (i.e. >80%) using a non-inferiority study design with 1-sided hypothesis testing (Farrington and Manning 1990) to determine whether or not the sensitivity of the EUS/EBUS diagnostic technique is inferior (i.e. 10% or more lower) when compared to the sensitivity of malignant mediastinal adenopathy of about 40%. This study requires subjects to agree to the selection of their standard of care procedure. Subjects will be randomized (stratified computer generated randomization stratified y center and y CT positivity for pathologically enlarged [>1cm short axis] node - 10 strata). Randomization will use variable block sizes (4-8), so that randomization allocation remains concealed as investigators will not be blinded. This study requires subjects to consent to the release of outcome data and follow-up data to be used for study analysis. No additional visit will be required for this study; this study will not require any additional time requirements beyond their scheduled evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or greater
* Pt is a surgical candidate for mediastinoscopy, thoracoscopy, or lung resection
* Known or suspected non-small cell carcinoma of the lung eligible for resection
* CT scan performed within 45 days prior to evaluation for study participation
* PET scan performed within 45 days prior to evaluation for study participation

Exclusion Criteria:

* Pathologically proven metastatic disease
* History of malignancy within 5 years other than (skin) basal cell carcinoma
* Enlarged ipsilateral mediastinal lymph nodes > 2.5 cm in diameter
* Peripheral T1 tumors with normal mediastinal lymph nodes on CT and PET

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Develop an integrated staging technique to detect early metastases in lung cancer which should affect patient outcomes more accurately than conventional staging techniques. | Post operative

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Hoffman, M.D., Study Chair — Medical University of South Carolina; Eric S Edell, M.D., Principal Investigator — Mayo Clinic, Rochester, MN; Michael Wallace, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina